CLINICAL TRIAL: NCT06378242
Title: An Single-arm, Multicenter Phase I/II Clinical Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Intravesical Instiliations of Disitamab Vedotin in Patients With High-risk Non-muscular Invasive Bladder Cancer (NMIBC) That Express HER2
Brief Title: To Evaluate the Safety, Efficacy, and Pharmacokinetics of Intravesical Instiliations of Disitamab Vedotin in Patients With High-risk Non-muscular Invasive Bladder Cancer (NMIBC) That Express HER2
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C029
Record Dates: First submitted 2024-04-12; First posted 2024-04-22 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: High-risk Non-muscle Invasive Bladder Cancer
Keywords: HER2-expression; High-risk non-muscle invasive bladder cancer; intravesical instiliations
MeSH Terms: interventions — disitamab vedotin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamab Vedotin Intravesical instiliations :Dose escalation cohort (Experimental): Participants will receive Disitamab Vedotin for injection Intravesical instiliations into the bladder for 1 hour, D1, once a week.
  Interventions: Drug: Disitamab Vedotin for injection

INTERVENTIONS:
Drug: Disitamab Vedotin for injection — Intravesical instiliations into the bladder
  Other Names: RC48

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and pharmacokinetics of intravesical instiliations of Disitamab Vedotin in patients with high-risk non-muscular invasive bladder cancer (NMIBC) that express HER2

DETAILED DESCRIPTION:
This is a single-arm, multicenter phase I/II clinical study to evaluate the safety, efficacy, and pharmacokinetics of intravesical instiliations of Disitamab Vedotin in patients with high-risk non-muscular invasive bladder cancer (NMIBC) that express HER2.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary consent to participate in the study and signed the informed consent form.
2. Male or female, age 18-75 years (including both).
3. Histologic confirmed non-muscle invasive bladder urothelial carcinoma (NMIBC), and the risk group met the high-risk (including very high-risk) group.

   Note: High-risk NMIBC is a high-grade / G3 tumor meeting any of the following:

   a.Carcinoma in situ (CIS) b. T1 stage c. diameter>3cm d.Multiple tumors, or recurrent tumors.
4. Absence of resectable disease（Ta and/or T1 disease） after transurethral resection (TURBT) procedures (residual CIS acceptable;
5. The urologist assessed that radical surgery for bladder cancer was not suitable or the subject refused radical surgery for bladder cancer.
6. Tumor tissue samples were detected by immunohistochemistry (IHC) to satisfy HER2 expression of 1+, 2+ or 3+.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
8. Adequate heart, bone marrow, liver, kidney and coagulation function

Exclusion Criteria:

* 1. Invasive bladder cancer (T2 and above) and / or with regional lymph node and distant metastasis.

  2. Combined urothelial carcinoma outside the bladder (i. e., urethra, ureter or renal pelvis).

  3. Any other antitumor therapy received within 4 weeks before study administration, .

  4 Subjects plan to undergo major surgery during the study or within 4 weeks before the first dose.

  5, Known allergic to DV and its components or to any excipients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2029-03-15 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity(DLT) (Phase I) | Approximately 21 days
Incidence of Adverse event (Phase I) | Approximately 1 years
  According to the NCI CTCAE V5.0, to evaluate safety including adverse event rate and adverse event grade
Recommended Phase II Dose(RP2D) | Approximately 21 days
  Assessed based on the Incidence of DLT
Maximum Tolerated Dosage(MTD) | Approximately 21 days
  Assessed based on the Incidence of DLT

SECONDARY OUTCOMES:
Disease-free survival (DFS) rates | Up to approximately 2 years
  Disease-free survival (DFS) rates was defined as the time from the date of first study treatment to the time of the subject's first high-grade Ta, T1 of any grade, CIS lasting greater than or equal to 6 months, new carcinoma in situ (CIS), cystectomy, disease progression, or death from any cause
Duration of response (DOR) | Up to approximately 2 years
  Defined as the time from the start of the first assessment of CR to the first assessment of high grade Ta, any grade of T1, new CIS, disease progression, cystectomy, or death from any cause
Disitamab Vedotin anti-drug antibody (ADA) | Up to approximately 2 years
  The number and proportion of anti-drug antibody (ADA)-positive subjects were analyzed according to dose group and time point.
PK of enfortumab vedotin: Maximum concentration (Cmax) | Approximately 1 years
  Cmax will be recorded from the PK blood samples collected.
PK of enfortumab vedotin: Trough concentration (Ctrough) | Approximately 1 year
  Ctrough will be recorded from the PK blood samples collected.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Sun Yat-sen Memorial Hospital,SunYat-sen University, Guangzhou, Guangdong
  - Tongji Hospital, Wuhan, Hubei
  - Hunan Cancer hospital, Changsha, Hunan
  - The first affiliated hospital with nanjing medical universtity, Nanjing, Jiangsu
  - West China Hospital, Chengdu, Sichuan
  - Tianjin Medical University Second Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Chen X, Huang M, Chen Z, Zhang C, Pan B, Liu C, Xu W, Fang J, Huang J, Lin T. Intravesical Disitamab Vedotin (RC48) for HER2-Expressing High-Risk Non-Muscle-Invasive Bladder Cancer: A Single-Arm, Dose-Escalation Phase I Trial Study. MedComm (2020). 2025 Jul 13;6(7):e70288. doi: 10.1002/mco2.70288. eCollection 2025 Jul. PMID 40661136